CLINICAL TRIAL: NCT06247189
Title: Onco-ICOPE: ICOPE Program Feasibility in the Management of Myeloma Patients Over 70 Years
Brief Title: ICOPE Program Feasibility in the Management of Myeloma Patients
Acronym: Onco-ICOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/22/0485
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Multiple Myeloma
Keywords: ICOPE; multiple myeloma; older patients; follow-up; frailty; geriatric nursing
MeSH Terms: conditions — Frailty; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICOPE Monitor Program (Experimental): Evaluation at inclusion and re-evaluation monthly.
  Interventions: Other: ICOPE Monitoring

INTERVENTIONS:
Other: ICOPE Monitoring — At inclusion set up of the ICOPE monitor program on the patient's device and evaluation (all steps) of ICOPE Monitor program.
  Monthly, re-evaluation of the patient (Step 1 and others if necessary ) according to the ICOPE Monitor program

SUMMARY:
This project proposes to adapt monthly the existing ICOPE (Integrated Care for Older People) MONITOR program for elderly myeloma patients. This adaptation aims to detect earlier functional decline and prevent loss of autonomy.

DETAILED DESCRIPTION:
With a median age of 70 years at diagnosis, multiple myeloma is a disease of the elderly, with 30-40% of patients over 75 years. Patients identified as frail have a higher risk of mortality, an increase in non-haematological adverse events and a significantly higher risk of treatment discontinuation. Comprehensive geriatric assessment is time-consuming, difficult to follow up regularly, and not routinely offered. However, this population presents an increased risk of loss of autonomy, linked both to age and treatment. For all seniors, ambition of ICOPE (Integrated Care for Older People) program is healthy aging by developing and maintaining their functional ability. To achieve this, the World Health Organization (WHO) recommends monitoring the evolution of intrinsic capacity, every 4 to 6 months. This covers 6 areas: mobility, memory, nutrition, psychological state, vision and hearing. This program is divided into 5 steps (Annex1). Adapting this monitoring to a monthly rhythm will prevent loss of autonomy in this population at greater risk. Early detection allows implementation of early and individualized care plan, thus limiting decline which could prove irreversible.

At inclusion, patient will be included in ICOPE MONITOR program. During this visit, the patient will undergo step 1 of the program, an evaluation of functional autonomy and quality of life, as well as a clinical examination and a collection of hematological data. If anomalies are detected, following steps (2-3-4-5) will be done.

Monthly, patient will carry out a screening (Step1) on his own. In case of abnormalities, following steps can be performed.

Visits will be made every 3 months with a screening (Step1), and if necessary, following steps, an evaluation of autonomy and an evaluation of quality of life.

Patients will be followed for 12 months. At the last visit the patient and the nurse will answer satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 70 years,
* Patient with multiple myeloma
* WHO performance status 0-3,
* Patient eligible for first- or second-line treatment
* Patient willing to participate in ICOPE MONITOR program
* Patient or caregiver able to use digital tools of ICOPE MONITOR: application or chatbot (computer or tablet or smartphone)
* Patient with a life expectancy of more than 3 months,
* Patient or caregiver able to understand, read and speak French
* Person affiliated or benefiting from a social security.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Patient in palliative care
* Patient participating in a study evaluating another frailty prevention program
* Patient unable to understand the study
* Patient under court protection, guardianship or curatorship,
* Patient refusal.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the implementation | 12 months
  Feasibility will be assessed on patient adherence to ICOPE MONITOR program. An interruption of 3 or more consecutive Step 1 over one year, apart from death, will be considered a failure of adherence for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BOURGADE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No